CLINICAL TRIAL: NCT05521633
Title: Comparison of the Effects of Metformin and Pioglitazone on Liver Enzymes
Brief Title: Comparison of the Effects of Metformin and Pioglitazone on Liver Enzymes and Ultrasound Changes in Non-Diabetic Non-Alcoholic Fatty Liver
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Mohammad Ibrahim, Postgraduate Resident of Internal Medicine, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: King EdwardMU
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Metformin; Pioglitazone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin Group (Active Comparator): Group-A; every participant took 500 mg of metformin daily
  Interventions: Drug: Metformin and Pioglitazone
- Pioglitazone Group (Active Comparator): Group-B; every participant took 30 mg of pioglitazone daily
  Interventions: Drug: Metformin and Pioglitazone

INTERVENTIONS:
Drug: Metformin and Pioglitazone — Every participant in Group-A took tablet metformin 500 mg daily and every participant in Group-B took tablet pioglitazone 30 mg daily.

SUMMARY:
BACKGROUND: Non-alcoholic fatty liver disease (NAFLD) is a spectrum of hepatic disease ranging from fat accumulation in liver to fibrosis and cirrhosis. It affects 25% of the world population on average. Objective of this study is to compare the effect of metformin (1000 milligrams daily) versus pioglitazone (30 milligrams daily) in improving liver transaminases and ultrasound changes in non-diabetic patients of NAFLD when given for six months.

METHODS: A Quasi-experimental study was conducted in Mayo Hospital Lahore from October 2019 to November 2020.Out of 96 half Patients were assigned randomly to Group-A (metformin) or Group-B (pioglitazone). Demographic history, abdominal ultrasound & liver enzymes were recorded on Proforma monthly till 6 months. Data was put into and analyzed by SPSS version 26; t-test was used to compare the mean liver transaminases between the two groups. Ultrasound findings were compared by Chi square. The P value of less than 0.05 was counted as significant.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Both male and female
2. Age: 18-80 Years
3. Ultrasound evidence of fatty liver as per operational definition
4. Liver enzymes as per operational definition

Exclusion Criteria:

1. Pregnancy
2. Cirrhotic patients as per operational definition
3. Chronic Hepatitis B or chronic hepatitis C
4. Patients taking long term steroids, highly active antiretroviral therapy, diltiazem, irinotecan, oxaliplatin and amiodarone
5. Patients taking alcohol (based on history and AST to ALT ratio)
6. Patients with heart failure (NYHA Classification class III or IV status: patients comfortable at rest but less than ordinary physical activity causes undue fatigue, dyspnea or palpitations)
7. Patients with renal failure (serum creatinine ≥ 1.4 mg% or eGFR < 45 ml/min/1.73 m2)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Liver transaminase levels | The comparison is done after 6 months of drug treatment
  There should be a 22% or more change in transaminases levels from baseline.

SECONDARY OUTCOMES:
Fatty Liver Grade | The comparison is done after 6 months of drug treatment
  There should be a change of liver fat content determined by ultrasound as Fatty Liver Grade

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mohammad Ibrahim, MBBS, MD, Principal Investigator — King Edward Medical University
Locations (1):
- King Edward Medical University/Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No